CLINICAL TRIAL: NCT06308458
Title: Effect Of The Breather Exerciser Trainer On Diaphragmatic Mobility And Thickness In Elderly
Brief Title: Breather Exerciser Trainer on Diaphragmatic Mobility And Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adly A Adam (Other)
Responsible Party: Sponsor-Investigator, Adly A Adam, Lecturer of Physical Therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003966
Record Dates: First submitted 2024-02-23; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Aging Well
Keywords: Breather Exerciser Trainer

STUDY DESIGN:
Intervention Model Description: Prospective pre/ posttreatment, randomized controlled study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double masking (Investigator, Outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (A) (Experimental): Experimental (Breather Exerciser Trainer + conventional breathing exercises) Group 30 healthy elders will receive inspiratory muscle training by breather exerciser trainer (Gradual intensity from 2-3 rate of perceived exertion (RPE) up to reach 5-7 RPE, with gradual frequency; 1st week 8 sets of 5 repetitions '1 minute rest', 2nd week be 9 sets, and 3rd week reach 10 sets of 5 repetitions. then from 4-8 weeks 'end of study protocol' will be 10 sets of 6 repetitions with 1 minute rest between sets.), along with conventional breathing exercises (Diaphragmatic breathing, Pursed-up breathing, and Exercise connected with respiration), for 5 sessions per week for eight weeks.
  Interventions: Other: Breather Exerciser Trainer; Other: Conventional Breathing Exercise
- Control Group (B) (Other): Control (conventional breathing exercises) Group:
  30 health elders will receive conventional breathing exercises (Diaphragmatic breathing; Pursed-up breathing, Exercise connected with respiration for 5 times a week for a total 8 weeks
  Interventions: Other: Conventional Breathing Exercise

INTERVENTIONS:
Other: Breather Exerciser Trainer — Gradual intensity from 2-3 rate of perceived exertion (RPE) up to reach 5-7 RPE, with gradual frequency; 1st week 8 sets of 5 repetitions '1 minute rest', 2nd week be 9 sets, and 3rd week reach 10 sets of 5 repetitions. then from 4-8 weeks 'end of study protocol' will be 10 sets of 6 repetitions with 1 minute rest between sets.), along with conventional breathing exercises (Diaphragmatic breathing, Pursed-up breathing, and Exercise connected with respiration), for 5 sessions per week for eight weeks
  Arms: Study Group (A)
Other: Conventional Breathing Exercise — Diaphragmatic breathing; place one hand on upper chest and the other on belly. Patient Breathe in slowly through nose, letting the air in deeply towards lower belly then patient is asked to tighten abdominal muscles and let them fall inward during exhalation through pursed lips Pursed-up breathing; by inhales through nose and exhales over 4 and 6 seconds in a whistling position Exercise connected with respiration; repetitive bilateral shoulder flexion then repetitive bilateral shoulder abduction, synchronized with breathing

SUMMARY:
The purpose of this study is to the effect of the breather exerciser trainer on diaphragmatic mobility and thickness in elderly.

DETAILED DESCRIPTION:
Egypt is the most populous country in Middle East, with expected elder population will reach 20.8% in 2050. Almost, old population undergo sarcopenia, and dynapenia including respiratory musculatures that may associated with elevated mortality rate. Such physiological deteriorations have a potential impact on the elders quality of life.

Therefore, regular specific breathing and exercise training may promote healthier life, and permits more mechanical efficient breathing pattern, thus older population could live a hassle-free life. older adults can maintain and improve their lung capacity.

ELIGIBILITY:
Inclusion Criteria:

* Age range 65-75 years old of both genders
* Oriented elder subjects assessed for cognitive impairment with score greater than 30 on Mini- Mental Scale.
* Healthy elders with normal pulmonary function test values according to reference values.

Exclusion Criteria:

* Using any medications affect muscular strength.
* Active hemoptysis, untreated pneumothorax, recent esophageal surgeries.
* Acute or chronic pulmonary diseases, or decompensated heart failure.
* Acute upper respiratory stenosis 'true vocal fold mass, vocal fold paralysis in adducted position, sub-glottic stenosis' or recent oral, facial or skull trauma or surgeries, also acute sinusitis, epistaxis, hemodynamic instability, tympanic membrane rupture, or acute middle ear pathology 'otitis or labyrinthitis'.
* Active smokers.
* Subjects with previous neurological disorders affecting respiratory muscles or any muscular dystrophies.
* Subjects with previous cervical or thoracic surgeries.
* Presence of hemodynamic instability 'heart rate more than 150beat per minute, or systolic blood pressure more than 140 mmHg, or diastolic blood pressure more than 90 mmHg'
* Presence of severe cognitive impairments affects their understanding of any steps of study protocol.
* Uncooperative individuals during chest ultrasound measurement that require performance of deep inspiration and full expiration.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickness in millimeters | Pretreatment and post treatment of 8 weeks of study protocol
  Preirus ultrasound device (Hitachi Medical Systems, Tokyo, Japan), with A 6-13 MHz linear probe will be utilized for diaphragm thickness assessment. Diaphragm thickness will be measured from the 8th or 9th intercostal space. Diaphragm thickness will measure thickness on expiration and during deep breathing to assess percentage of thickening during inspiration. and diaphragm thickness will expressed in millimeters.
Diaphragmatic mobility in centimeters | pretreatment and post treatment of 8 weeks of study protocol
  Preirus ultrasound device (Hitachi Medical Systems, Tokyo, Japan). a 1-5 MHz convex probe will be used for diaphragm mobility assessment. Diaphragm mobility will be measured from the costal line junction of the medial axillary line. The excursions of two hemidiaphragms will be measured using two-dimensional or M-mode ultrasonography, during respiratory maneuvers. Diaphragmatic mobility will be expressed in centimeters.

SECONDARY OUTCOMES:
Functional Capacity | pretreatment and post treatment of 8 weeks of study protocol
  Will use Six-Minute Walk Test, as a self-paced submaximal field exercise test to determine functional capacity according to standard procedures administrated in a 30 meters hallway.
Geriatric Quality of life Questionnaire | pretreatment and post treatment of 8 weeks of study protocol
  Will use Quality of Life Questionnaire to assess functional disability and evaluate quality of life through a comprehensive geriatric 15-dimensional standardized, self-administrated measure for health-related quality of life questionnaire. The single index score (item of 15 dimensions) on a 1-5scale, representing the overall quality of life, is calculated from the health state descriptive system by using a set of population-based preference or utility weights.
  Best quality of life score is 15 'best quality of life- it is the lowest score could gained' that means sum all included items score of 1 referring to best quality of life for each dimension of the questionnaire.
  While worst sum value is 75 'worst- highest score could gained, as in complete bedridden' that refers to each subitem score was 5.
Geriatric Quality of Life | pretreatment and post treatment of 8 weeks of study protocol
  Will use Katz Questionnaire as a suitable tool for assessing functional status and capability to perform activities of daily living independently.
  Where 0 is the lowest score refers to complete dependent person. While 6 is the highest score refers to independent person.

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen G El Nahas, PHD, Study Chair — Head of department and Professor of Cardiovascular, Respiratory disorders, Geriatric Department; Samir A El Gazar, PHD, Study Director — Head of department and Professor of Cardiovascular, Respiratory disorders, Geriatric Department; Donia M El-Masry, MSc, Principal Investigator — Lecturer of Physical Therapy for Cardiovascular, Respiratory disorders and Geriatric
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study purpose, Selection, and randomization, detailed intervention procedures, and statistical analysis, plus revealed results and conclusion
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3-5months
Access Criteria: adampt80a@gmail.com